CLINICAL TRIAL: NCT03344133
Title: Effect of a 4-week Moderate Intensity Exercise Programme on Gut Microbiota, Cardiovascular Disease Risk Factors and Appetite Regulation in Overweight Women
Brief Title: Effect of Exercise Programme on Gut Microbiota, CVD Risk Factors and Appetite Regulation in Overweight Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Konstantinos Gerasimidis, Senior Lecturer, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 200140132
Record Dates: First submitted 2017-09-19; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Overweight and Obesity
Keywords: Obesity; Exercise; CVD risk factors; Appetite Regulation; Gut Microbiota
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): 4-week moderate intensity exercise programme
  Interventions: Behavioral: Exercise
- Control (No Intervention): 4 weeks of habitual life style

INTERVENTIONS:
Behavioral: Exercise — 4-week moderate intensity exercise programme
  Arms: Exercise

SUMMARY:
Evidence suggests that gut microbiota contributes to the development of atherosclerosis and therefore CVDs. Exercise has been extensively reported to be protective against CVDs due to modification of body fatness, metabolic risk factors and cardio-respiratory fitness. It remains unclear whether impact of exercise on CVD risk can be at least in part explained by changes in the microbiota. It also remains to be investigated whether modification of appetite and appetite hormones due to participation in exercise are related to changes in the gut microbiota composition. Therefore, this study will be conducted in overweight, healthy, sedentary women and will investigate the effect of a 4-week moderate intensity exercise programme on gut microbiota composition and metabolic activity, plasma concentrations of fasting and postprandial lipids, glucose, insulin and inflammatory markers, fasting and postprandial gut appetite hormones, subjective appetite measures and cardio-respiratory fitness.

DETAILED DESCRIPTION:
Study Design: This is a randomized controlled study with a parallel design. Healthy, sedentary females aged between 18-45 years old will be recruited by means of an advertisement leaflet and word of mouth. Eligible participants will be enrolled in the study and will be randomly allocated to either exercise intervention (EX) or control (C) groups. The EX group will participate in a 4-week exercise intervention and the C group will be asked to continue with habitual life style for 4 weeks. Before and after 4 weeks of the intervention, participants from both groups will be asked to conduct a submaximal exercise test and a 7-hour experimental trial during which blood samples will be collected and metabolic rate will measured before and after consumption of standardized breakfast and lunch. Prior to the first 7-hour trial, participants will be asked to record diet for 3 days and replicate this diet prior to the second 7-hour trial. During these 3 days participants will provide fresh stool samples. Participants allocated to control group will have the option to participate in exercise intervention. A subset of the participants will repeat a 7-hour experimental trial and provide fresh stool and urine sample after 7 days of detraining.

Methods:

Preliminary Health Check: Participants will undertake a health screening questionnaire on the day of recruitment. Participants will also need to fill in Physical Activity Readiness Questionnaire (PARQ). Only participants who answered "no" to all questions in PARQ will conduct the submaximal exercise test.

Anthropometry: All participants will have height, weight and waist circumference measured at baseline and 4 weeks after the intervention.

7-hour Experimental Trial: Participants will attend the metabolic suite (New Lister Building, Glasgow Royal infirmary) in a fasted state at approximately 9.00 am. Participants will be instructed to lie supine on the couch, with the head resting on the pillow provided. Resting metabolic rate will be measured for 20 minutes and fasting blood sample will be obtained. A breakfast meal will be consumed immediately after the fasting sample and a lunch meal after 4 hours. Blood samples will be taken throughout a cannula hourly after breakfast and lunch consumption. Following each blood sample, metabolic rate will be measured for the duration of 20 minutes. Prior each blood sample, participants will fill in appetite questionnaires. Blood samples will be analysed for plasma lipids, glucose, insulin, inflammatory markers and gut appetite hormones using standard existing procedures.

Feacal sample collection & analysis: A disposable stool sample collection kit will be provided prior to the 7-hour trial day. Once collected, the container is sealed and placed in a larger sealable bag with a reducing sachet to remove oxygen and maintain anaerobic bacteria. Stool samples will be measured for changes in gut microbiota based on 16S rRNA amplicon sequencing, bacterial functional capacity and targeted bacterial metabolites (short chain fatty acids, sulphide, ammonia).

Exercise Training Programme: Exercise training will consist of 4 weekly sessions of endurance type exercise (cycling and running) lasting for 30, 40, 50, 60 minutes in the week 1, 2, 3 and 4 respectively. The time and day of each training trial will be agreed between the investigator and the participant and will be based around the participant's availability. All exercise sessions will be supervised by a researcher.

Submaximal Exercise Test: Participants will exercise on treadmill at gradually increasing intensities until 85% of maximal heart rate. During the last minute of each of the intensities heart rate will be measured and expired air will be collected by Douglas bag technique and analysed for oxygen consumption and carbon dioxide production. Relation between heart rate and rate of oxygen consumption will be used to predict maximal oxygen consumption, a marker of cardio-respiratory fitness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, sedentary females, BMI>25 kg/m2, on a stable body weight for the last 3 months

Exclusion Criteria:

* Acute or chronic illness, use of antibiotics the past 3 months, smoking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2015-09-16 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota composition | 12 months
  Changes in the gut microbiota composition measured by 16S rRNA amplicon sequencing.

SECONDARY OUTCOMES:
Interleukin-6 (IL-6) | 3 months
  Changes in fasting and postprandial interleukin-6 pre- and post-interventions measured by Human IL-6 ELISA Ready-Set-Go (Affymetrix, eBioscience)
Glucose | 3 months
  Changes in fasting glucose pre- and post-interventions measured by Randox Glucose
Triglycerides | 3 months
  Changes in fasting and postprandial triglycerides pre- and post-interventions measured by Randox Triglycerides
Insulin | 3 months
  Changes in fasting insulin pre- and post-interventions measured by Mercodia Insulin ELISA
Peptide YY (PYY) | 12 months
  Changes in fasting and postprandial peptide YY pre- and post-interventions measured by Human PYY (Total) ELISA (Merc Millipore)
Glucagon-like peptide-1 (GLP-1) | 12 months
  Changes in fasting and postprandial glucagon-like peptide-1 pre- and post-interventions measured by GLP-1 Total ELISA (Merc Millipore)
Subjective appetite | 12 months
  Changes in subjective appetite (hunger, satiety, fullness, prospective food consumption, desire to eat) pre- and post-interventions measured by Visual Analogue Scales (VAS) where respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points (minimum score is 0 and maximum score is 100)
Faecal short-chain fatty acids | 12 months
  Changes in concentrations of feacal short-chain fatty acids pre- and post-interventions measured by TRACE 2000 Gas Chromatography (ThermoQuest Ltd)
Faecal pH | 1 month
  Changes in feacal pH between pre- and post-intervention measured by Hanna HI 98140
Body weight | 1 month
  Differences in body weight (kilograms) between pre- and post-intervention measured by TANITA scales (TBF-300)
Height | 1 month
  Height (meters) measured by stadiometer, a vertical ruler with a sliding horizontal paddle which is adjusted to rest on the top of the head
Body fat (kilograms) | 1 month
  Differences in body fat expressed in kilograms between pre- and post-intervention measured by TANITA scales (TBF-300)
Body fat (% percentage) | 1 month
  Differences in body fat expressed as percentage (%) (proportion of fat to the total body weight) between pre- and post-intervention measured by TANITA scales (TBF-300)
Body Mass Index (BMI) | 1 month
  Differences in body mass index (weight and height will be combined to report BMI in kg/m^2) between pre- and post-intervention measured by TANITA scales (TBF-300)
Dietary Intake | 6 months
  Energy intake and macro nutrient intake using WinDiets software based on food composition tables
Maximum Oxygen Consumption | 2 weeks
  Maximum Oxygen Consumption (ml/kg/min) measured before and after the interventions by Servomex Gas Analyser
Energy substrate oxidation | 6 months
  Fat and carbohydrate oxidation in the fasted and postprandial state measured before and after the interventions using indirect calorimetry (Oxycon Pro)
Resting Metabolic Rate | 2 month
  Resting metabolic rate was measured before and after the interventions (Oxycon Pro)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Gerasimidis, BSc MSc PhD, Principal Investigator — University of Glasgow
Locations (1):
- School of Medicine, University of Glasgow / New Lister Building, Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No